CLINICAL TRIAL: NCT05038592
Title: Phase I/II Study of Tagraxofusp in Combination With Decitabine for Patients With Myelomonocytic/Myeloproliferative Neoplasm and High Risk Myelodysplastic Syndromes
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0895; NCI-2021-04293 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0895 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-01; First posted 2021-09-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia; Chronic Myelomonocytic Leukemia-1; Chronic Myelomonocytic Leukemia-2; Myelodysplastic/Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic-Myeloproliferative Diseases | interventions — Decitabine; Injections; tagraxofusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, tagraxofusp-erzs) (Experimental): Patients receive decitabine IV over 60 minutes on days 1-5, and tagraxofusp-erzs IV over 15 minutes on days 1-3. Cycles of decitabine repeat every 28 days in the absence of disease progression or unacceptable toxicity. Treatment with tagraxofusp-erzs repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Tagraxofusp-erzs

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Biological: Tagraxofusp-erzs — Given IV
  Other Names: Diphtheria Toxin(388)-Interleukin-3 Fusion Protein; DT(388)-IL3 Fusion Protein; DT388IL3 fusion protein; Elzonris; IL3R-targeting Fusion Protein SL-401; SL-401; Tagraxofusp; Tagraxofusp ERZS

SUMMARY:
This phase I/II trial studies the side effects, best dose, and effect of tagraxofusp and decitabine in treating patients with chronic myelomonocytic leukemia. Tagraxofusp consists of human interleukin 3 (IL3) linked to a toxic agent called DT388. IL3 attaches to IL3 receptor positive cancer cells in a targeted way and delivers DT388 to kill them. Chemotherapy drugs, such as decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving tagraxofusp and decitabine may help to control the disease in patients with chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability and maximum tolerable dose (MTD) of tagraxofusp-erzs (tagraxofusp) in combination with decitabine.

II. To assess overall response (OR) rate to tagraxofusp in combination with decitabine.

SECONDARY OBJECTIVES:

I. To assess overall survival (OS), duration of response, relapse-free survival (RFS) and safety profile.

II. Correlative studies.

OUTLINE: This is a phase I, dose-escalation study of tagraxofusp-erzs followed by a phase II study.

Patients receive decitabine intravenously (IV) over 60 minutes on days 1-5, and tagraxofusp-erzs IV over 15 minutes on days 1-3. Cycles of decitabine repeat every 28 days in the absence of disease progression or unacceptable toxicity. Treatment with tagraxofusp-erzs repeats every 28 days for up to 7 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The participant is ≥ 18 years old
* Diagnosis of myelodysplastic/myeloproliferative neoplasm (MDS/MPN) according to World Health Organization (WHO) and:

  * Phase 1 dose escalation portion: CMML-1 or CMML-2 by WHO or higher-risk MDS (defined as IPSS-Revised score >3.5 or with TP53 mutations) with >5% blasts or MDS/MPN (other than CMML) with >5% bone marrow blasts and no response after 6 cycles of azacitidine, decitabine, guadecitabine or ASTX727 (decitabine-cedazuridine) or relapse or progression after any number of cycles
  * Phase 2 dose expansion portion:

    * Relapsed cohort (Cohort A): CMML-1 or CMML-2 or higher-risk MDS (defined as IPSS-Revised score >3.5 or with TP53 mutations) with >5% blasts or MDS/MPN (other than CMML) with >5% bone marrow blasts by WHO and no response after 6 cycles of azacitidine, decitabine, guadecitabine or ASTX727 (decitabine-cedazuridine) or relapse or progression after any number of cycles
    * Hypomethylating agents (HMA) naive cohort (Cohort B): previously untreated CMML-1 or CMML-2 and intermediate-2 or high-risk IPSS or higher-risk MDS (defined as IPSS-Revised score >3.5 or with TP53 mutations) with >5% blasts or MDS/MPN (other than CMML) with >5% bone marrow blasts.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2
* Left ventricular ejection fraction (LVEF) ≥ 50% as measured by multigated acquisition scan or 2-dimensional (2-D) echocardiogram (ECHO) within 28 days prior to start of therapy and no clinically significant abnormalities on a 12-lead electrocardiogram (ECG)
* Serum creatinine ≤ 1.5 mg/dL (or ≤ 114 umol/L)
* Serum albumin ≥ 3.2 g/dL (or ≥ 32 g/L) in the absence of receipt of (IV) albumin within the previous 72 hours
* Total Bilirubin =< 1.5 mg/dL (or ≤ 26 umol/L)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN)
* Creatine kinase (CK) ≤ 2.5 times the ULN
* If a woman of child bearing potential (WOCBP), the participant has a negative serum or urine pregnancy test within 1 week prior to tagraxofusp treatment (intervals shorter than 1 week are acceptable, if required by institutional guidelines).
* The participant has signed informed consent prior to initiation of any study-specific procedures or treatment.
* The participant is able to adhere to the study visit schedule and other protocol requirements, including follow-up for response assessments.
* The participant (either male or female) agrees to use acceptable contraceptive methods for the duration of time in the study, and to continue to use acceptable contraceptive methods for 2 months after the last tagraxofusp infusion.

Exclusion Criteria:

* Participants has persistent clinically significant toxicities Grade .2 from previous chemotherapy not readily controlled by supportive measures (excluding alopecia, nausea, and fatigue).
* Participants has received treatment with chemotherapy, wide-field radiation, or biologic therapy within 14 days of study entry.
* Participants has received treatment with another investigational agent within 14 days of study entry or concurrent treatment with another investigational agent.
* Participants has previously received treatment with tagraxofusp or has a known hypersensitivity to any components of the drug product.
* Participants has an active malignancy and/or cancer history (excluding myeloproliferative disorders and concomitant myeloid malignancies as specified in the inclusion criteria) that is requiring active therapy. Participants with the following neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including superficial bladder cancer), cervical intraepithelial neoplasia, or organ- confined prostate cancer with no evidence of progressive disease.
* Participants has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina, or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
* Participants has uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that, in the Investigator's opinion, would put the patient at significant risk for pulmonary complications during the study.
* Participants has known active or suspected disease involvement of the central nervous system (CNS). If suspected due to clinical findings, CNS disease should be ruled out with relevant imaging and/or examination of cerebrospinal fluid.
* Participants is receiving immunosuppressive therapy, with the exception of corticosteroids (maximum dose of 10 mg prednisone or equivalent) and tacrolimus for prophylaxis of graft-versus-host disease (GVHD). If the patient has been on immunosuppressive treatment for active GVHD, the treatment(s) for active GVHD must have been discontinued at least 14 days prior to study drug and there must be no evidence of Grade .2 GVHD.
* Participants has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness that would limit compliance with study requirements.
* Participants is pregnant or breast feeding.
* Participants has known human immunodeficiency virus (HIV).
* Participants has evidence of active or chronic Hepatitis B or Hepatitis C infection.
* Participants is oxygen-dependent.
* Participants has any medical condition that in the Investigator's opinion place the patient at an unacceptably high risk for toxicities.
* Hydroxyurea is permitted only in settings in which a patient had been receiving this agent prior to study entry; hydroxyurea may only be administered during Cycle 1. After Cycle 1, the use of hydroxyurea may be permitted in consultation with the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2027-01-29 (Estimated); Study Completion 2027-01-29 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose (Phase I) | At end of cycle 1 (1 cycle = 28 days)
Incidence of dose limiting toxicities (Phase I) | Up to end of cycle 1 (1 cycle = 28 days)
Overall response (OR) (Phase II) | After 2 cycles of therapy (1 cycle = 28 days)
  Will estimate the OR for the combination treatment along with the 95% credible interval. The association between OR rate and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M Bravo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org